# **Cover Page**

Project RESIST: Increasing Resistance to Tobacco Marketing Among Young Adult Sexual Minority Women Using Inoculation Message Approaches

NCT04812795

Date Oct 11 2021

### UNIVERSITY OF PENNSYLVANIA RESEARCH SUBJECT INFORMED CONSENT FORM

**Protocol Title:** Project RESIST – Increasing resistance to Tobacco Marketing

Among Young Adult Sexual Minority Women Using

Inoculation Message Approaches

Principal Investigator:

Andy Tan, PhD, MPH, MBA, MBBS

## **Key Information**

### Introduction

We are inviting you to take part in a research study. Research is a way of gaining new knowledge. A person who participates in a research study is called a "participant." This research study is evaluating various marketing strategies that may be used in health interventions designed to reach sexual minority women.

It is expected that about 2000 people will take part in this research study.

An institution that is supporting a research study either by giving money or supplying something that is important for the research is called the "sponsor." The sponsor of this protocol is the National Cancer Institute and is providing the funding for this study.

This research consent form explains why this research study is being done, what is involved in participating in the research study, the possible risks and benefits of participation, alternatives to participation, and your rights as a research participant. The decision to participate is yours. If you decide to participate, please select "Yes, I consent" at the end of the form. You have the option to download a copy so that you can refer to it while you are involved in this research study.

## What should I know about a research study?

- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

# Why is this research being done?

This research is being done to test the effectiveness of images, symbols, and language for health messaging about reducing cigarette smoking. We will show you several images and ask you questions about those images to assess their effectiveness.

## How long will I take part in this research?

This initial survey will take approximately 20 minutes and you will be asked to complete a follow up survey of about 20 minutes in one month. Additionally, we will be sending you weekly health messages which will take less than a minute to view.

More detailed information about the study procedures can be found under the "How long will I be in this research study?" section if you request additional information.

## Is there any way being in this study could be bad for me?

There is no physical risk. There is minimal psychological risk. There is low risk to your privacy.

More detailed information about the risks of this study can be found under the "What are the risks and discomforts of this research study?" section if you request additional information.

## Will being in this study help me in any way?

There are no direct benefits to you from your participation in this research. We cannot promise any benefits to others from your participation in this research. However, possible benefits to others may include the development of more effective health messages.

# Will I be compensated for being in this study?

Yes, you will be paid according to the description of the study and breakdown by Prolific's requirements

## What happens if I do not want to be in this research?

Your alternative to participating in this research study is to not participate.

By selecting "Yes, I agree to participate," I acknowledge:

- I have had enough time to read the consent and think about participating in this study;
- I am willing to participate in this study;
- I understand my participation is voluntary and I can withdraw at any time
- Yes, I agree to participate
- No, I do not wish to participate
- I would like more information

### **Detailed Information**

#### A. <u>Introduction</u>

We are inviting you to take part in a research study. Research is a way of gaining new knowledge. A person who participates in a research study is called a "participant." This research study is evaluating various marketing strategies that may be used in health interventions designed to reach sexual minority women.

It is expected that about 2000 people will take part in this research study.

An institution that is supporting a research study either by giving money or supplying something that is important for the research is called the "sponsor." The sponsor of this protocol is the National Cancer Institute and is providing the funding for this study.

This research consent form explains why this research study is being done, what is involved in participating in the research study, the possible risks and benefits of participation, alternatives to participation, and your rights as a research participant. The decision to participate is yours. If you decide to participate, please select "Yes, I consent" at the end of the form. You have the option to download a copy so that you can refer to it while you are involved in this research study.

#### B. WHY IS THIS RESEARCH STUDY BEING DONE?

This research is being done to test the effectiveness of images, symbols, and language for health messaging about reducing cigarette smoking. We will show you several images and ask you questions about those images to assess their effectiveness.

#### C. WHAT OTHER OPTIONS ARE THERE?

Taking part in this research study is voluntary. You can decide not to participate in this research study

#### D. WHAT IS INVOLVED IN THE RESEARCH STUDY?

This research study involves the completion of this survey, which will take approximately 20 minutes. During the baseline survey, you will be randomly assigned to one of two study groups. After the baseline survey, you will receive 5 additional health messages over email in 1, 2 and 3 weeks. Finally, you will be asked to complete a follow up survey in one month, which takes about 20 minutes.

#### E. HOW LONG WILL I BE IN THIS RESEARCH STUDY?

This initial survey will take approximately 20 minutes and you will be asked to complete a follow up survey of about 20 minutes in one month. Each weekly health message should take you less than a minute to view.

In addition, you can stop participating in the research study at any time.

#### F. WHAT ARE THE RISKS OR DISCOMFORTS OF THE RESEARCH STUDY?

There are risks to taking part in any research study.

- Physical risks: There are no physical risks to participating in this study.
- Psychological risks: The risk of participation is minimal. You will be asked to view anti-smoking messages and tobacco ads. Viewing of these publicly available ads is not expected to be different from everyday viewing of advertisements. There is minimal risk of psychological distress when completing certain sensitive risk questions within the survey.
- Privacy risks: The risks to privacy are very low. We do not ask for any personally identifiable data. We ensure that your data is protected through data confidentiality procedures as well.

To reduce the risk to participating in this study, please note that you may choose not to enroll and you can skip any question that you do not wish to answer.

#### G. WHAT ARE THE BENEFITS OF THE RESEARCH STUDY?

There are no direct benefits of the research to participants. We hope the information learned from this research study will provide more information about the effectiveness of advertising images targeted towards minority groups.

#### H. CAN I STOP BEING IN THE RESEARCH STUDY AND WHAT ARE MY RIGHTS?

You have the right to choose not to sign this form. If you decide not to sign this form, you cannot participate in this research study.

You can stop being in the research study at any time, by exiting the survey or closing the window.

If you choose to not participate, or if you are not eligible to participate, or if you withdraw from this research study, this will not cause any penalty or loss of benefits to which you are otherwise entitled.

#### I. WHAT ARE THE COSTS?

There are no costs to you for participating.

#### J. WHAT ABOUT CONFIDENTIALITY?

We will take measures to protect the privacy and security of all your personal information, but we cannot guarantee complete confidentiality of study data.

The study team plans to publish the results of this research study and when we do, we may be asked to share the data we collect available to other researchers. We will not include information that identifies you in any publications or to the researchers who request the data to do research.

This study may be registered on <a href="https://www.clinicaltrials.gov">https://www.clinicaltrials.gov</a>, a publicly available registry of clinical trials. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### K. WHOM DO I CONTACT IF I HAVE QUESTIONS ABOUT THE RESEARCH STUDY?

If you have questions, concerns or complaints regarding your participation in this research study or if you have any questions about your rights as a research subject, you should speak with Andy Tan by phone (215-746-6546) or email: andy.tan@asc.upenn.edu If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the IRB at (215) 898 2614.

#### L. FUTURE USE OF DATA

Your personal information collected during this study may be stored and used for future research. If so, any personal identifiers will be removed so that the information cannot be linked back to you. As a result, we will no longer be able to identify you through the data.

Investigators, including investigators from collaborating institutions, can request this data for new research. De-identified data may also be shared with outside non-profit academic investigators as well as with non-profit LGBT-serving organizations.

You will not be asked to provide additional informed consent for the use of your deidentified information in future research.

### M. **DOCUMENTATION OF CONSENT**

By selecting "Yes, I agree to participate," I acknowledge:

- I have had enough time to read the consent and think about participating in this study;
- I am willing to participate in this study;
- I understand that my participation is voluntary and I can withdraw at any time
- Yes, I agree to participate
- No, I do not wish to participate